CLINICAL TRIAL: NCT00622999
Title: Effects of Malnutrition on Colon Cancer Patients With Abdominal Surgery
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Dr. med. Zeno Sanga, Inselspital Bern
Other Study IDs: Malnutr_Colon_CH_2007; Study ID: 2000/049
Record Dates: First submitted 2008-02-14; First posted 2008-02-25 (Estimated); Last update posted 2011-03-11 (Estimated); Status verified 2011-03

CONDITIONS: Malnutrition; Colon Cancer
Keywords: Malnutrition; Colon cancer; Colon surgery; Outcome; Complication rate
MeSH Terms: conditions — Malnutrition; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All: All patients

SUMMARY:
The prevalence of malnutrition in patients with colorectal cancer is recorded. We want to find out, if a malnourished patient has more complications after the elective surgery.

DETAILED DESCRIPTION:
All patients attending elective colorectal surgery are screened for malnutrition in advance. Their length of stay in the hospital and the complications are recorded.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal Carcinoma
* Elective surgery
* Informed consent

Exclusion Criteria:

* Survival < 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing colorectal surgery with diagnosed malignity.
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2003-01; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Complication rate | during stay

SECONDARY OUTCOMES:
Mortality | during stay

CONTACTS AND LOCATIONS:
Overall Officials: Stefan F Mühlebach, Prof, Study Chair — Kantonsspital Aarau, Switzerland
Locations (1):
- Kantonsspital, Aarau, Switzerland